CLINICAL TRIAL: NCT00453765
Title: Prospective Single-centre, Double Blind Randomised Trial of Montelukast in Patients With Chronic Cough and Bronchial Hyperreactivity
Brief Title: The Effect of Montelukast in Patients With Chronic Cough and Bronchial Hyperreactivity
Acronym: montelukast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Jan W.K. van den Berg, Dr., Isala
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL14828.075.06
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Cough; Bronchial Hyperreactivity
Keywords: cough; hyperreactivity; montelukast
MeSH Terms: conditions — Cough; Bronchial Hyperreactivity | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): montelukast
  Interventions: Drug: montelukast
- B (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast — montelukast, 8 weeks, once daily, 10 milligrams
  Other Names: singulair
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
The purpose is to determine whether montelukast during 6 weeks has superior antitussive effects (measured with the LCQ) compared with placebo in patients with cough lasting > 8 weeks and enhanced bronchial hyperreactivity.

DETAILED DESCRIPTION:
Chronic cough is a frequent problem in general practice and one of the most common reasons for referral to a respiratory clinic. Prospective studies have shown that the vast majority of cases of chronic cough are due to one or more of three conditions: rhinitis/postnasal drip syndrome, asthma and gastro-oesophageal reflux disease. Other significant causes of chronic cough include postviral (post-infectious) cough, and eosinophilic bronchitis. In only a minority of the patients with a chronic cough no cause can be found. This is called idiopathic cough.

Analysis and treatment of patients with chronic cough often proved to be difficult and disappointing. Nevertheless, centers in which a comprehensive diagnostic and therapeutic protocol was implemented reported excellent results. Therefore the first cough clinic is started in The Isala Klinieken, Zwolle/The Netherlands in 2004.

Asthmatic cough is often accompanied by the more typical symptoms of dyspnoea and wheezing. In a subgroup of asthmatics, however, cough is the sole or predominant symptom. This condition is termed cough-variant asthma (CVA). Cough due to CVA usually improves within the first week of inhaled bronchodilator therapy, however, complete resolution of cough may require up to 8 weeks of combination therapy with inhaled bronchodilators and corticosteroids. A subgroup of CVA patients with severe, refractory cough may require systemic (oral) steroids, alone or followed by inhaled therapy.

Leukotrienes are contributing significantly to the pathobiology of asthma. These 'pathways of asthma' could be suppressed by leukotriene inhibitors. Multiple clinical trials have demonstrated the ability of the leukotriene modifiers to improve symptoms, pulmonary function and bronchial hyperresponsiveness in chronic asthma, as well as in exercise-induced and aspirin-induced asthma. Until recently, the antitussive effects of this drug class had not been investigated properly. Spector and Tan concluded in a pilot trial with only 14 patients that 10 mg montelukast seems to be effective in CVA. However, nowadays in care of asthma, montelukast is widely used in a dosage of 10 mg. Therefore we intend to study the effects of montelukast on chronic cough (VAS-cough-score) on a wider patient population; is montelukast superior to placebo in the treatment of patients with chronic cough and a demonstrated bronchial hyperreactivity?

Aim of the study:

The purpose is to determine whether montelukast during 6 weeks has superior antitussive effects (measured with the VAS cough) compared with placebo in patients with cough lasting > 8 weeks and enhanced bronchial hyperreactivity.

Study design:

Montelukast trial: prospective single-centre, double blind randomised trial.

In the montelukast study 84 patients between 18 and 90 years old, referred to the cough outpatient clinic with chronic cough and enhanced bronchial hyperreactivity will be recruited after informed consent is obtained.

Patients will be randomised (for gender, age, smoking, duration of symptoms and the use of inhaled corticosteroids) to 6- week treatment with 10 mg daily montelukast or placebo. Before randomisation all patients have to fill in the Visual Analogue Scale (VAS) for detection of the degree of cough in the last 24 hours and the dutch version of the Leicester Cough Questionnaire (LCQ) for the detection of illness specific quality of life. Adverse events will be noted in this period. Finally, both groups will be compared.

Inhaled corticosteroids may be continued during the study at a constant dose. Nasal, ophthalmologic and dermatological steroids are allowed according to individual needs, but their dose should be kept constant throughout the trial.

H1 blockers, nasal anticholinergics as well as nasal or ophthalmologic preparations of nedocromil or cromoglycate are permitted for treatment of allergic rhinitis.

Study population:

Patients between 18 and 90 years old, referred to the cough outpatient clinic with chronic cough and enhanced bronchial hyperreactivity.

Intervention:

Patients between 16 and 90 years old, referred to the cough outpatient clinic with chronic cough and enhanced bronchial hyperreactivity will receive daily montelukast 10 mg or placebo during 6 weeks.

Main study endpoint :

1. Difference in cough VAS scores; montelukast vs placebo.

Secondary study endpoints:

1. Difference in average score on the Leicester Cough Questionaire (LCQ) between the two treatment groups; montelukast vs placebo.
2. Comparison of the adverse events of montelukast vs placebo.

Randomisation:

Patients will be randomised by a computer minimisation program for the following factors: gender, age, smoking, duration of symptoms and the use of inhaled corticosteroids.

Statistical analysis:

The primary analysis will be on an intention-to-treat basis. The mean change in the primary endpoint (LCQ total and domain scores) after 6 weeks between the groups will be analysed using an unpaired t-test. This test will also be used to analyse differences after 6 weeks in secondary endpoints (VAS cough score).

Since both the primary and secondary endpoints in the study will be measured more than two times (repeatedly measured) the course of these scores over time will be tested using MANOVA-analysis. To test for differences in proportions (proportion of patients with adverse events) the Chi2 -test will be used. Data analyses will be performed using SPSS version 12.

Burden, risks and advantages associated with participation:

Side effects have been reported in 10 % of the cases; mostly of headache and abdominal pain. Also gastrointestinal problems, allergic reactions, psychiatric disorders, liver, and haematological disorders could occur.

Interactions: Montelukast is metabolised by CYP3A4. Concomitant use of CYP3A4 inducing medication like fenytoïne, phenobarbital, or rifampicin must be prevented.

Medication metabolised by CYP2C8 must also be avoided, because in vitro studies have shown that montelukast is an powerful CYP2C8 inhibitor.

Benefits: superior resolution of cough compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 90 years old, referred to the cough outpatient clinic with chronic cough and enhanced bronchial hyperreactivity.
* chronic cough is defined as a cough > 8 weeks duration.
* enhanced bronchial hyperreactivity is a PD20 < 2.5 mg methacholine.

Exclusion Criteria:

* concomitant severe disease; lung cancer and diseases with a short life expectancy (< 1 year).
* patients suffering from COPD and/or other relevant lung diseases.
* clinically relevant abnormal laboratory values suggesting an unknown disease requiring further clinical evaluation.
* use of systemic steroids 4 weeks (injectable depot steroids 6 weeks) before entry into the baseline period, or more than 3 courses during the last 6 months.
* pregnancy.
* abnormal chest X-ray.
* use of medication inducing CYP3A4 (for example; fenytoïne, phenobarbital or rifampicin.
* use of medication metabolised by CYP2C8.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2007-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Difference in average score on the Leicester Cough Questionnaire (LCQ) between the two treatment groups; montelukast vs placebo. | 2 years

SECONDARY OUTCOMES:
Difference in cough VAS scores; montelukast vs placebo. | 2 years
Comparison of the adverse events of montelukast vs placebo. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Van Den Berg, MD, Study Director — Departement of Pulmonology
Locations (1):
- Isala Klinieken, Zwolle, Netherlands